CLINICAL TRIAL: NCT00319553
Title: Comparison in US Adolescents of the Safety and Immunogenicity of Two Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis (Tdap) Vaccines: ADACEL™ and BOOSTRIX®
Brief Title: Post-licensure, Modified Double-blind, Multi-center Study Evaluating Safety and Immunogenicity of ADACEL® and BOOSTRIX®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Td516
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Pertussis; Tetanus; Diphtheria
Keywords: Tetanus; diphtheria; acellular pertussis
MeSH Terms: conditions — Whooping Cough; Tetanus; Diphtheria | interventions — adacel; Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adacel® Vaccine Group (Experimental)
  Interventions: Biological: ADACEL®:Tetanus, Reduced Diphtheria and Acellular Pertussis Adsorbed
- BOOSTRIX® Vaccine Group (Active Comparator)
  Interventions: Biological: BOOSTRIX®: Tetanus, Reduced Diphtheria and Acellular Pertussis Adsorbed

INTERVENTIONS:
Biological: ADACEL®:Tetanus, Reduced Diphtheria and Acellular Pertussis Adsorbed — 0.5 mL, IM
  Other Names: ADACEL®
  Arms: Adacel® Vaccine Group
Biological: BOOSTRIX®: Tetanus, Reduced Diphtheria and Acellular Pertussis Adsorbed — 0.5 mL, IM
  Other Names: BOOSTRIX®
  Arms: BOOSTRIX® Vaccine Group

SUMMARY:
This is a descriptive study to evaluate the safety and immunogenicity of ADACEL® and BOOSTRIX® vaccines among US adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 - 18 years of age at the time of vaccination in this trial
* Signed Institutional Review Board (IRB)-approved informed assent / consent form.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a female, negative serum/urine pregnancy test.

Exclusion Criteria:

* Any condition which, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Serious chronic disease (i.e. cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric etc) that is unstable or that might:

  * interfere with the ability to participate fully in the study; or
  * interfere with evaluation of the vaccine.
* Known or suspected impairment of immunologic function.
* Febrile illness within the last 72 hours or an oral temperature ≥ 100.4°F (≥ 38°C) at the time of inclusion.
* History of documented tetanus, diphtheria or pertussis disease within the preceding 5 years.
* Known or suspected receipt of a tetanus or diphtheria-containing vaccine within the preceding 2 years.
* Known or suspected receipt of a pertussis-containing vaccine within the preceding 5 years.
* Administration of immune globulin or other blood products within the last three months, or injected or oral corticosteroids or other therapy expected to materially alter immune function within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting less than 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Received any vaccine in the 21-day period prior to enrollment or scheduled to receive any vaccination after enrollment and prior to visit 2.
* Suspected or known hypersensitivity to any of the vaccine components or to latex.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 647 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (9):
- United States (9):
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Frederick, Maryland
  - Durham, North Carolina
  - Franklin, Tennessee
  - Bellevue, Washington
  - Mercer Island, Washington
  - Sammamish, Washington
  - Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 09 May 2006 to 02 October 2006 in 12 clinical centers in the US.
Pre-assignment Details: A total of 647 participants who met the inclusion and exclusion criteria were enrolled, 644 were vaccinated and included in the analysis.
Period: Overall Study
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group
Started | 323 | 321
Completed | 319 | 317
Not Completed | 4 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group | Total
Number analyzed (Participants) | 323 | 321 | 644
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 291 | 291 | 582
  Between 18 and 65 years | 32 | 30 | 62
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.5 (2.33) | 14.7 (2.33) | 14.6 (2.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 150 | 304
  Male | 169 | 171 | 340
Region of Enrollment [Number; unit: participants]
  United States | 323 | 321 | 644

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting A Solicited Injection Site or Systemic Reactions Within 7 Days Following Vaccination With Adacel® or Boostrix®
Description: Solicited injection site reactions: Pain, Erythema, and swelling. Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia.
  Grade 3 reaction definitions: Pain = Incapacitating, unable to perform usual activities; Erythema and swelling = ≥ 5 cm; Fever = temperature ≥ 39.1°C or ≥ 102.3°F; Headache, Malaise, and Myalgia = Prevents daily activities.
Time Frame: Day 0 to 7 post-vaccination
Population: Solicited injection site and Systemic reactions were analyzed in the intent-to-treat safety population
Measure: Number; unit: Participants
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group
Number analyzed (Participants) | 320 | 317
Participants
  Any solicited injection site reaction | 273 | 257
  Grade 3 solicited injection site reaction | 5 | 4
  Any solicited injection site Pain | 270 | 247
  Grade 3 solicited inj. site Pain (Incapacitating) | 2 | 3
  Any solicited injection site Erythema | 75 | 67
  Grade 3 solicited injection site Erythema (≥ 5 cm) | 2 | 1
  Any solicited injection site Swelling | 61 | 44
  Grade 3 solicited injection site Swelling (≥ 5 cm) | 2 | 1
  Any solicited systemic reaction | 216 | 205
  Grade 3 solicited systemic reaction | 9 | 9
  Any solicited Fever | 18 | 9
  Grade 3 solicited Fever (≥ 39.1°C or ≥ 102.3°F) | 1 | 0
  Any solicited Headache | 136 | 108
  Gr 3 solicited Headache: Prevents daily activities | 3 | 4
  Any solicited Malaise | 91 | 78
  Gr 3 solicited Malaise: Prevents daily activities | 8 | 6
  Any solicited Myalgia | 167 | 166
  Gr 3 solicited Myalgia: Prevents daily activities | 1 | 3

2. Primary Outcome: Percentage of Participants With Tetanus Antitoxin Concentrations ≥ 0.1 IU/mL Pre- and Post-Vaccination With Adacel® or Boostrix®.
Time Frame: Day 0 and 28 days post-vaccination
Population: Tetanus antitoxin concentrations were analyzed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group
Number analyzed (Participants) | 305 | 304
Percentage of Participants
  Tetanus IgG antitoxin ≥0.1 IU/mL :pre-vaccination | 99 | 98
  Tetanus IgG antitoxin ≥0.1 IU/mL :28 days post-vac | 100 | 100

3. Primary Outcome: Percentage of Participants With Diphtheria Antitoxin Concentrations ≥ 0.1 IU/mL Pre- and Post-Vaccination With Adacel® or Boostrix®.
Time Frame: Day 0 and 28 days post-vaccination
Population: Diphtheria antitoxin concentrations were analyzed in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group
Number analyzed (Participants) | 305 | 304
Percentage of Participants
  Diphtheria IgG antitoxin ≥0.1 IU/mL : pre-vacc | 92 | 93
  Diphtheria IgG antitoxin ≥0.1 IU/mL: 28 D post-vac | 100 | 100

4. Primary Outcome: Geometric Mean Concentration of Antibody to Pertussis Antigens Pre- and Post-Vaccination With Adacel® or Boostrix®.
Time Frame: Day 0 and 28 days post-vaccination
Population: Geometric mean concentration of antibody to the pertussis antigens were analyzed in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group
Number analyzed (Participants) | 305 | 304
EU/mL
  Anti-pertussis toxoid IgG: pre-vaccination | 14.4 [12.5 to 16.6] | 13.5 [11.6 to 15.8]
  Anti-filamentous hemagglutinin IgG:pre-vaccination | 26.1 [22.7 to 30.0] | 28.2 [24.5 to 32.4]
  Anti-pertactin IgG: pre-vaccination | 12.4 [10.6 to 14.6] | 13.1 [11.2 to 15.5]
  Anti-fimbriae types 2 and 3 IgG: pre-vaccination | 13.9 [12.0 to 16.2] | 14.5 [12.2 to 17.2]
  Anti-pertussis toxoid IgG: post-vaccination | 86.7 [78.8 to 95.4] | 135.9 [122.9 to 150.2]
  Anti-filamentous hemagglutinin IgG post-vaccinat. | 240.7 [217.7 to 266.1] | 402.9 [365.5 to 444.2]
  Anti-pertactin IgG: post-vaccination | 322.7 [279.7 to 372.4] | 463.3 [395.4 to 542.9]
  Anti-fimbriae types 2 and 3 IgG: post-vaccination | 1203 [1004 to 1442] | 26.6 [22.2 to 31.8]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination up to 1 month post-vaccination.
Arm/Group | Adacel® Vaccine Group | Boostrix® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/323 | 0/321
Other Adverse Events (participants affected / at risk) | 273/320 | 257/317
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Adacel® Vaccine Group (N=320) | Boostrix® Vaccine Group (N=317)
Solicited injection site Pain (General disorders) | 270 | 257
Solicited injection site Erythema (General disorders) | 75 | 67/316
Solicited injection site Swelling (General disorders) | 61 | 44/316
Solicited Fever (General disorders) | 18 | 9/316
Solicited Headache (Nervous system disorders) | 136 | 108
Solicited Malaise (General disorders) | 91 | 78
Solicited Myalgia (Musculoskeletal and connective tissue disorders) | 167 | 166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.